CLINICAL TRIAL: NCT04689984
Title: The Benefits of Astaxanthin as Add on Therapy in the Management of Painful Diabetic Neuropathy Patient: Randomized Clinical Trial
Brief Title: The Benefits of Astaxanthin as Add on Therapy in the Management of Painful Diabetic Neuropathy Patient
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duta Wacana Christian University (Other)
Collaborators: PT SOHO Global Health Tbk (Unknown)
Responsible Party: Principal Investigator, Rizaldy Taslim Pinzon, Principal investigator, Neurologist, Duta Wacana Christian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASTAXANTHIN
Record Dates: First submitted 2020-12-19; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Astaxanthin; Standard therapy; Neuropathy; Diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Standard of Care; astaxanthine

STUDY DESIGN:
Intervention Model Description: Eligible subjects were randomly allocated to receive any of the following regiments: standard therapy consists of pregabalin, gabapentine, or amitriptyline (control group) or standard therapy and astaxanthin 6 mg tablet once daily (experimental group).
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Receive standard therapy consists of gabapentin, pregabalin, or amitriptyline and astaxanthin 6 mg tablet once daily (experimental group).
  Interventions: Drug: Standard therapy; Drug: Astaxanthin
- Control Group (Active Comparator): Receive standard therapy consists of gabapentin, pregabalin, or amitriptyline.
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Standard therapy — Gabapentin, pregabalin, or amitriptyline
Drug: Astaxanthin — Astaxanthin 6 mg tablet once daily
  Arms: Experimental Group

SUMMARY:
Diabetes is one of the main health care problemsworldwide with 5% average increased number of cases every year. According to International Diabetes Federation the prevalence of people with diabetes reached the number of 425 million people in 2017 and estimated rising to 628 million by 2045. Painful Diabetic Neuropathy (PDN) is the most common complication of diabetes affecting 90% of the patients. The symptoms of PDN include numbness, burning, stabbing pain, paraesthesia or hyperesthesiaof both symmetrical limbthat could reduce the quality of life. Several studies have found several therapeutic options to cope with pain in the PDN, but the results are not as satisfactory due to the uncertain pathophysiology of the disease and the limitations of the drug that can be administered because of itspolypharmaceutical side effects. The causes of diabetic neuropathy not only include vascular and metabolic factors but also Reactive Oxygen Species.

There are several therapeutic options that can be administered such as glycemic index arrangement,foot care, symptomatic treatment, and predominantly pain therapy. According to guidelines, there are drugs therapy thatrecommended for PDN, among others, Gabapentin, Pregabalin and anticonvulsants until the pain subsides. Unfortunately, this treatment is only aimed at relieving the symptoms of existing pain but not working on existing pathophysiological mechanisms and fixing sensory deficits of neuropathy trials. Multi-target treatments is needed to attenuate neuronal inflammation, oxidative stress and apoptosis. Additional therapy can be an option to support healing and also the process of metabolic pathophysiology that occurs due to rising glycemic index in the body that causes the work of hexosamine pathway and trigger the formation of ROS and inflammation. There is evidence of research demonstrating the neuroprotective effects of Astaxanthin as oxidative, anti-inflammatory and anti-apoptotic agent. Not only that, Astaxanthin is also a good supplement addition with no toxic effects when consumed, as well as hydrophilic and also lipophilic nature which makes Astaxanthin can penetrate the BBB effectively.

DETAILED DESCRIPTION:
Detailed Description:

This was randomized clinical trial, active comparator, open label, controlled study from the period of November 2020 - November 2021 at Bethesda Hospital, Yogyakarta, Indonesia.

There were 60 painful diabetic neuropathy patients who fulfilled the inclusion and exclusion criteria. Each subject had been followed up from the first day of medication administration until 8 weeks after medication administration.

Ethical approval number ((kosong)) was obtained from Health Research Ethics Committee, Bethesda Hospital Yogyakarta.

The hypothesis of this study:

a. Add on oral astaxanthin to standard treatment in patients with painful diabetic neuropathy is more effective in reducing pain and neuropathic symptoms in 8 weeks of treatment compared with standard treatment, b. Add on oral astaxanthin to standard treatment in patients with painful diabetic neuropathy is as safe as standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Adult age (>18 years old)
* Diagnosed as painful diabetic neuropathy based on validated Diabetic Neuropathy Symptoms (DNS) and Diabetic Neuropathy Examination (DNE)

Exclusion Criteria:

* Subjects with significant renal and liver problem
* Subjects with known hypersensitivity to astaxanthin
* Pregnancy and breastfeeding patients
* Patients that enrolled any clinical trial within a month
* Not competent enough in giving approval and answering questionnaires

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Improvement in Visual Analogue Scale (VAS) at week 4 | 4 weeks after treatment initiation
  Change in pain impact on daily life as measured by Visual Analogue Scale (VAS) from its baseline value. Visual analogue scale is a continuous scale comprised of a horizontal or vertical line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100). The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Improvement in Visual Analogue Scale (VAS) at week 8 | 8 weeks after treatment initiation
  Change in pain impact on daily life as measured by Visual Analogue Scale (VAS) from its baseline and week 4 value. Visual analogue scale is a continuous scale comprised of a horizontal or vertical line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100). The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Improvement in Numeric Pain Scale at week 4 | 4 weeks after treatment initiation
  Change in pain impact on daily life as measured by Numeric Pain Scale from its baseline value. Numeric pain scale is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. Higher scores indicating greater pain intensity.
Improvement in Numeric Pain Scale at week 8 | 8 weeks after treatment initiation
  Change in pain impact on daily life as measured by Numeric Pain Scale from its baseline and week 4 value. Numeric pain scale is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. Higher scores indicating greater pain intensity.
Improvement in Brief Pain inventory at week 4 | 4 weeks after treatment initiation
  Change in pain impact on daily life as measured by Brief Pain Inventory from its baseline value. The Brief Pain Inventory evaluates a patient's pain experience through a number of different scales. There are line drawings of the front and back of a human body on which patients mark the location of their pain. Patients are asked to list the treatments or medications that they are using and how much relief they have provided in the past 24 hours. In addition, patients fill out 11 different numeric rating scale that ask about pain intensity (ranging from 0 to 10) and the effect of the pain on their ability to function during various activities of daily living. A higher score indicates greater pain intensity.
Improvement in Brief Pain inventory at week 8 | 8 weeks after treatment initiation
  Change in pain impact on daily life as measured by Brief Pain Inventory from its baseline and week 4 value. The Brief Pain Inventory evaluates a patient's pain experience through a number of different scales. There are line drawings of the front and back of a human body on which patients mark the location of their pain. Patients are asked to list the treatments or medications that they are using and how much relief they have provided in the past 24 hours. In addition, patients fill out 11 different numeric rating scale that ask about pain intensity (ranging from 0 to 10) and the effect of the pain on their ability to function during various activities of daily living. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Rizaldy T Pinzon, MD, MSc, PhD, Principal Investigator — Duta Wacana Christian University
Locations (1):
- Bethesda Hospital Yogyakarta, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fakhri S, Aneva IY, Farzaei MH, Sobarzo-Sanchez E. The Neuroprotective Effects of Astaxanthin: Therapeutic Targets and Clinical Perspective. Molecules. 2019 Jul 20;24(14):2640. doi: 10.3390/molecules24142640. PMID 31330843
- [Background] Iqbal Z, Azmi S, Yadav R, Ferdousi M, Kumar M, Cuthbertson DJ, Lim J, Malik RA, Alam U. Diabetic Peripheral Neuropathy: Epidemiology, Diagnosis, and Pharmacotherapy. Clin Ther. 2018 Jun;40(6):828-849. doi: 10.1016/j.clinthera.2018.04.001. Epub 2018 Apr 30. PMID 29709457
- [Background] Javed S, Alam U, Malik RA. Treating Diabetic Neuropathy: Present Strategies and Emerging Solutions. Rev Diabet Stud. 2015 Spring-Summer;12(1-2):63-83. doi: 10.1900/RDS.2015.12.63. Epub 2015 Aug 10. PMID 26676662
- [Background] Juster-Switlyk K, Smith AG. Updates in diabetic peripheral neuropathy. F1000Res. 2016 Apr 25;5:F1000 Faculty Rev-738. doi: 10.12688/f1000research.7898.1. eCollection 2016. PMID 27158461
- [Background] Kaur S, Pandhi P, Dutta P. Painful diabetic neuropathy: an update. Ann Neurosci. 2011 Oct;18(4):168-75. doi: 10.5214/ans.0972-7531.1118409. PMID 25205950
- [Background] Rosenberger DC, Blechschmidt V, Timmerman H, Wolff A, Treede RD. Challenges of neuropathic pain: focus on diabetic neuropathy. J Neural Transm (Vienna). 2020 Apr;127(4):589-624. doi: 10.1007/s00702-020-02145-7. Epub 2020 Feb 8. PMID 32036431
- [Background] Schreiber AK, Nones CF, Reis RC, Chichorro JG, Cunha JM. Diabetic neuropathic pain: Physiopathology and treatment. World J Diabetes. 2015 Apr 15;6(3):432-44. doi: 10.4239/wjd.v6.i3.432. PMID 25897354
- [Background] Snyder MJ, Gibbs LM, Lindsay TJ. Treating Painful Diabetic Peripheral Neuropathy: An Update. Am Fam Physician. 2016 Aug 1;94(3):227-34. PMID 27479625
- [Background] Wu H, Niu H, Shao A, Wu C, Dixon BJ, Zhang J, Yang S, Wang Y. Astaxanthin as a Potential Neuroprotective Agent for Neurological Diseases. Mar Drugs. 2015 Sep 11;13(9):5750-66. doi: 10.3390/md13095750. PMID 26378548